CLINICAL TRIAL: NCT05350020
Title: An Open Label Pilot Study to Investigate the Effects of Two Preparations of Hydrocortisone (Hydrocortisone 100mg/ml and Solu-Cortef) Injected Intramuscularly Into the Deltoid and Upper Thigh Muscle During the State of Hypocortisolaemia
Brief Title: The Effects of Two Brands of Hydrocortisone Injected Intramuscularly Into Deltoid and Thigh Muscles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The London Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ATC 017
Record Dates: First submitted 2022-03-29; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Addison's Disease
MeSH Terms: conditions — Addison Disease | interventions — hydrocortisone hemisuccinate; Injections; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Solu-Cortef® in deltoid muscle (Experimental): Solu-Cortef® in deltoid muscle
  Interventions: Drug: Solu-Cortef 100 MG Injection
- Solu-Cortef® in thigh muscle (Experimental): Solu-Cortef® in thigh muscle
  Interventions: Drug: Solu-Cortef 100 MG Injection
- Hydrocortisone 100mg/ml in deltoid muscle (Experimental): Hydrocortisone 100mg/ml in deltoid muscle
  Interventions: Drug: Hydrocortisone 100mg/ml
- Hydrocortisone 100mg/ml in thigh muscle (Experimental): Hydrocortisone 100mg/ml in thigh muscle
  Interventions: Drug: Hydrocortisone 100mg/ml

INTERVENTIONS:
Drug: Solu-Cortef 100 MG Injection — Licensed medicine used in clinical practice. Preparations will be used unmodified in this trial withinmarketing authorisations.
  Arms: Solu-Cortef® in deltoid muscle; Solu-Cortef® in thigh muscle
Drug: Hydrocortisone 100mg/ml — Licensed medicine used in clinical practice. Preparations will be used unmodified in this trial within marketing authorisations.
  Arms: Hydrocortisone 100mg/ml in deltoid muscle; Hydrocortisone 100mg/ml in thigh muscle

SUMMARY:
The study will be looking at the cortisol profiles of hypocortisolaemic patients following 100mg injections of two hydrocortisone preparations (Solu-Cortef® & Hydrocortisone 100mg/ml). The investigators plan to use two methods of intramuscular injection to administer the preparations, one using a 1inch orange needle into the deltoid muscle and the other using a 1.25inch blue needle into the thigh muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 inclusive
2. Written informed consent provided, prior to any study related assessments/procedure being conducted.
3. Men & Women with a BMI between 18-30kg/m2
4. Addison's disease or Bilateral Adrenalectomised patients with pre-hydrocortisone cortisol level below 100nmol/L and ACTH greater than 50ng/L on screening visit
5. All patients must be stabilised on hydrocortisone with no change in dosage for 6 months, other than transient increases for concurrent illness.
6. Able to self-inject into deltoid and thigh muscles following teaching at recruitment.
7. Female patients of child-bearing potential must be willing to use an acceptable method of birth control/abstinence from the time consent is signed until 6 weeks after treatment is discontinued. Acceptable methods include: physical barrier (male or female condom, contraceptive sponges, diaphragms and cervical caps),-contraceptive pill or patch, spermicidal method alongside a physical barrier or an intrauterine device (IUD). Abstinence is also acceptable if it falls in line with the patient's usual lifestyle however it must be complete abstinence and not either; periodic, ovulation timed, symptothermal or withdrawal based. Those patients that utilise hormonal contraceptives must have used the same method for at least three months before additional barrier contraception (as described above). Patients of non-child-bearing potential are defined as having 12 month amenorrhoea or are surgically sterile.

Exclusion Criteria:

1. Patient on oestrogen based or mixed oral contraceptives unless willing to use alternate effective method of contraception
2. Patient on any forms of oral steroids other than hydrocortisone.
3. Any patient with secondary adrenal failure
4. Patients with a diagnosis of any disease or condition listed in Hydrocortisone 100mg/ml and Solu-Cortef®'s SmPC as being contraindicated or precautionary for use
5. Patient with concurrent illness in the week preceding screening/study visit.
6. Patient must not have had an adrenal crisis in the week before screening
7. Patient with Nelson's syndrome.
8. Participating in another IMP investigation
9. Patient who is unable or unwilling to comply with the protocol.
10. Patient taking any medications/substances that are known to interact with hydrocortisone e.g. CYP3A4 inhibitors
11. Pregnant or breastfeeding patients
12. Patient has any other disease or condition that, in the opinion of the investigator, might compromise patient safety or interfere with the results of the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
State of Hypocortisolaemia when injected into deltoid muscle or thigh muscle | 4 weeks
  Measure of Peak Serum Cortisol

SECONDARY OUTCOMES:
Pain perception following use of difference sizes of needles (1inch orange needle versus 1.25inch blue needle), muscle groups (deltoid versus thigh) and hydrocortisone preparations (Solu-Cortef® versus Hydrocortisone 100mg/ml) | 4 Weeks
  Verbal Numerical Rating Scale for Pain from 0 (no pain) to 10 (worst pain) Size of needle Injection site used Hydrocortisone preparation
Hydrocortisone absorption | 4 Weeks
  Measured by Injection site circumference measured in Centimeters and BMI (weight in kilograms, height in meters) BMI combined to view Area under curve and Time to peak concentration
Ability to Self-Inject | 4 Weeks
  Measure by assessment of the following: Hypocortisolaemia symptoms Leftover IMP in ampoules (Quanitity of IMP measure in ml to calculate remaining mg of IMP) Time taken to inject
Subjective health status/impact on quality of life | 5 Weeks
  AddiQol score (AddiQol Health-related quality of life in Addison's disease) total score 30 Ability to self-inject

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Bouloux, Principal Investigator — Endocrinology Consultant
Locations (1):
- The London Clinic, London, United Kingdom